CLINICAL TRIAL: NCT02509000
Title: Beijing Indoor Air Purifier Intervention Study
Acronym: BIAPSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WeiHuang (Other)
Collaborators: Peking University Third Hospital (Other); Utrecht University (Other)
Responsible Party: Sponsor-Investigator, WeiHuang, Peking University School of Public Health, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: WHuang14
Record Dates: First submitted 2015-07-20; First posted 2015-07-27 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-07

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active-mode (Active Comparator): Air purifier in active-mode
  Interventions: Other: air purifier
- Sham-mode (Sham Comparator): Air purifier in sham-mode
  Interventions: Other: air purifier

INTERVENTIONS:
Other: air purifier — filtration units randomly allocated to active- and sham-mode in 20 recruited households for four weeks

SUMMARY:
This study aimed to assess the impact of air filtration on indoor air quality and cardio-pulmonary health in residents living in high outdoor pollution settings in Beijing.

ELIGIBILITY:
Inclusion Criteria:

* Global Initiative for Chronic Obstructive Lung Disease criteria (mild to moderate, GOLD stage I~II;
* severe to very severe, GOLD stage III~IV) quit smoking for at least 1 year;
* a ratio of pre-bronchodilator forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) equal to or less than 0.70 and an increase of FEV1 with the use of 400μg of albuterol of less than 12% of the pre-bronchodilator one;
* no history of asthma or any other active lung disease.
* Subjects were free from exacerbations for at least 6 weeks.

Exclusion Criteria:

* Patients with heart pacemaker,
* heart failure with bundle-branch block,
* recent myocardial infarction (in the last 12 weeks) and
* anticoagulant therapy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
respiratory inflammation | 4 weeks
  analyzed EBC pH and inflammation biomarkers 8-isoprostane and nitrite and nitrate

SECONDARY OUTCOMES:
systemic inflammation | 4 weeks
  analyzed systemic inflammation biomarkers C-reaction Protein, Blood coagulation factor fibrinogen (Fib), Interleukin (IL) -8, -1β, -6, -10, -12p70 and tumor necrosis factor-α (TNF-α)
oxidative stress | 4 weeks
  analyzed systemic oxidative stress biomarker urinary 8-hydroxy-2-deoxyguanosine (8-OHdG)

OTHER OUTCOMES:
lung function | 4 weeks
  lung function test (FEV1, FEV1 %predicted, FEV1/FVC, 176 maximum midexpiratory flow (MMEF), MMEF %predicted) using an Aspirometer
autonomic function | 4 weeks
  twelve-hour ambulatory electrocardiogram (ECG) and blood pressure (BP) were monitored

CONTACTS AND LOCATIONS:
Overall Officials: Wei Huang, PhD, Principal Investigator — Peking University School of Public Health